CLINICAL TRIAL: NCT06721988
Title: Exploring the Effect of Preventive Analgesia with Oxycodone and Parecoxib Sodium on the Chronification of Acute Pain in Adult Patients Underwent Laparoscopic-assisted Abdominal Major Surgery
Brief Title: Effect of Preventive Analgesia with Oxycodone and Parecoxib Sodium on the Chronification of Acute Post-operative Pain
Acronym: AOPC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ailin Luo (Other)
Collaborators: Jinhua Central Hospital (Other); Minda Hospital of Hubei Minzu University (Unknown); Taihe Hospital of Traditional Chinese Medicine (Unknown); Qujing first people's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Ailin Luo, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TJ-IRB202411042
Record Dates: First submitted 2024-11-27; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Oxycodone; Chronic Pain, Postoperative
Keywords: Oxycodone; Preventive analgesia; Chronification of acute postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OP group (Experimental): Participants in this group will receive oxycodone and parecoxib sodium before surgical incision.
  Interventions: Drug: oxycodone and parecoxib sodium combinations
- PP group (Placebo Comparator): Participants in this group will receive a placebo and parecoxib sodium before surgical incision.
  Interventions: Drug: Placebo and parecoxib sodium combinations

INTERVENTIONS:
Drug: oxycodone and parecoxib sodium combinations — Participants will receive 0.1ml/kg oxycodone (1mg/ml) and 2 ml parecoxib sodium (20 mg/ml) combinations after the anesthesia induction but before the surgical incision. Oxycodone is administered 5 minutes after parecoxib sodium administration.
  Arms: OP group
Drug: Placebo and parecoxib sodium combinations — Participants will receive 0.1ml/kg placebo (0.9% saline) and 2 ml parecoxib sodium (20 mg/ml) combinations after the anesthesia induction but before the surgical incision. Placebo is administered 5 minutes after parecoxib sodium administration.
  Arms: PP group

SUMMARY:
The goal of this clinical trial is to learn if the administration of oxycodone for preventive analgesia works to reduce the chronification of acute postoperative pain in adult participants undergoing major abdominal surgery. The main question it aims to answer is:

• Does administration of oxycodone before surgical incision reduce the occurrence of chronic pain or relieve the chronic pain symptoms 3 months after the operation? Researchers will compare oxycodone + parecoxib sodium to placebo + parecoxib sodium combinations to see if oxycodone works to reduce the chronification of acute postoperative pain.

Participants will:

* Take oxycodone + parecoxib sodium or placebo + parecoxib sodium combinations before the surgical incision
* Cooperate with the follow-up staffs and complete some checkups or tests within 3 months after the operation.

DETAILED DESCRIPTION:
Preventive analgesia encompasses a range of analgesic strategies designed to mitigate hyperalgesia and allodynia induced by noxious stimuli by preventing peripheral and intraoperative sensitization to pain. It constitutes a fundamental component of multimodal analgesia. Nonsteroidal anti-inflammatory drugs (NSAIDs) are presently the most frequently employed agents for preventive analgesia, demonstrating efficacy in reducing the incidence of acute postoperative pain and chronic post-surgical pain. However, the management of acute postoperative pain and chronic post-surgical pain remains suboptimal. κ-opioid receptors are regarded as the primary receptors involved in the transmission of visceral pain, and κ-receptor agonists have been shown to effectively inhibit this transmission. Administering κ-receptor agonists via intravenous infusion either before the conclusion of surgery or postoperatively can substantially mitigate pain during the recovery period. This indicates that κ-receptor agonists possess potential as preventive analgesics. However, there is currently a paucity of high-quality clinical evidence supporting their use in preventive analgesia. Oxycodone functions as a dual agonist of μ-opioid and κ-opioid receptors and is extensively utilized in postoperative analgesia and anesthesia induction. Its safety and efficacy in pain management have been thoroughly validated. Theoretically, the concurrent administration of oxycodone and NSAIDs, which mitigate pain signal transmission through distinct mechanisms, could result in an additive preventive analgesic effect. However, there is currently a paucity of high-quality clinical evidence supporting this hypothesis. Consequently, this study seeks to investigate the effects of the combined administration of oxycodone and NSAIDs as preventive analgesia on the transition of acute postoperative pain to chronic pain in patients undergoing major abdominal surgery. The findings aim to contribute clinical evidence and theoretical insights to enhance perioperative pain management strategies.

ELIGIBILITY:
Inclusion Criteria:

* ASA I~III；
* BMI ranging from 18 to 28 kg/m²；
* For elective laparoscopic-assisted major abdominal surgery under general anesthesia;
* Estimated surgical duration (from incision to the last suture of the skin) was at least 2 hours.

Exclusion Criteria:

* Pregnant or lactating patients;
* Patients diagnosed with septic shock or multiple organ failure within 14 days;
* Patients with preoperative severe electrolyte disorders;
* Patients with stroke, transient ischemic attack, or other similar events within the past 3 months
* Patients with unstable angina, myocardial infarction within the past 3 months; or presence of untreated arrhythmia or arrhythmia not well-controlled with treatment;
* Patients with diabetes, uncontrolled blood glucose levels, or diabetes complications such as diabetic ketoacidosis, hyperosmolar coma, diabetes-related infections, diabetic nephropathy, retinopathy, diabetic cardiomyopathy, diabetic peripheral neuropathy, diabetic foot, etc. before the surgery;
* Patients with severe liver dysfunction (Child-Pugh score > 6), renal dysfunction (GFR < 90 ml/(min•1.73m²));
* Exploratory surgeries, day surgeries, or surgeries that only involve opening and closing the abdomen;
* Blood pressure ≥180/110 mmHg at rest (≥Grade 3 hypertension according to the 2020 ISH Hypertension Guidelines); or systolic blood pressure <90 mmHg or mean blood pressure <65 mmHg;
* Patients participated in other drug trials within the past 3 months;
* Patients with communication difficulties, inability to understand pain scores or patient-controlled intravenous analgesia;
* Patients with consciousness disorders or other psychiatric illnesses;
* Patients with a confirmed or suspected history of substance abuse or long-term use of anesthetic sedatives and analgesics;
* Cancer patients have received neoadjuvant treatment or chemotherapy preoperatively;
* Allergic to the drugs used in this trial and their components.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1316 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Visceral pain scores in the surgical area at 90 days postoperatively. | 90 days after the surgery
  The pain scores will be assessed by the Numeric Rating Scale (NRS) and Brief Pain Inventory Scale-Short form (BPI-9). The NRS evaluates pain intensity on a 0-10 scale and the scores are grouped as no (NRS 0), mild (NRS 1-4), moderate (NRS 5-7), or severe pain (NRS 8-10). The BPI-9 is a 9-item questionnaire and each item is scored from 0 = no pain to 10 = worst pain. The BPI-9 is used to assess various aspects of pain severity and pain interference.
The incidence of moderate to severe visceral pain at 90 days postoperatively. | 90 days after the surgery
  The incidence will be calculated as the ratio of the number of participants with moderate to severe visceral pain to the number of participants allocated to each group at 90 days after the surgery .

SECONDARY OUTCOMES:
Somatic pain scores in the surgical area at 48 hours postoperatively; | 48 hours after the surgery
  The pain scores will be assessed by the NRS and BPI-9 scales as described above.
Visceral pain scores in the surgical area at 48 hours postoperatively; | 48 hours after the surgery
  The pain scores will be assessed by the NRS and BPI-9 scales as described above.
Incidence of moderate to severe visceral pain at 48 hours postoperatively; | 48 hours after the surgery
  The incidence will be calculated as the ratio of the number of participants with moderate to severe visceral pain to the number of participants allocated to each group at 48 hours after the surgery.
Incidence of moderate to severe visceral pain in the surgical area at 30 days postoperatively; | 30 days after the surgery
  The incidence will be calculated as the ratio of the number of participants with moderate to severe visceral pain to the number of participants allocated to each group at 30 days after the surgery.
Incidence of moderate to severe somatic pain in the surgical area at 30 days postoperatively; | 30 days after the surgery
  The incidence will be calculated as the ratio of the number of participants with moderate to severe somatic pain to the number of participants allocated to each group at 30 days after the surgery.
Incidence of moderate to severe somatic pain in the surgical area at 90 days postoperatively. | 90 days after the surgery
  The incidence will be calculated as the ratio of the number of participants with moderate to severe somatic pain to the number of participants allocated to each group at 90 days after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Ailin, Principal Investigator — Department of Anesthesiology of Tongji hospital

IPD SHARING:
Plan to Share IPD: No